CLINICAL TRIAL: NCT06079398
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Placebo-controlled Trial, Evaluating Safety, Tolerability, and Efficacy of Subcutaneous Doses of TransCon CNP Administered Once Weekly for 52 Weeks in Infants (0 to <2 Years of Age) With Achondroplasia Followed by an Open Label Extension (OLE) Period
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of TransCon CNP Compared With Placebo in Infants (0 to <2 Years of Age) With Achondroplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASND0030
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Navepegritide (Experimental): Once weekly double-blinded treatment with SC injection of 100 µg/kg of Navepegritide for 52 weeks
  Interventions: Drug: Navepegritide
- Placebo for Navepegritide (Placebo Comparator): Once weekly double-blinded treatment with SC injection of 100 µg/kg of Placebo for Navepegritide for 52 weeks
  Interventions: Drug: Placebo for Navepegritide

INTERVENTIONS:
Drug: Navepegritide — Once-weekly subcutaneous injection of 100 µg/kg Navepegritide
  Arms: Navepegritide
Drug: Placebo for Navepegritide — Once-weekly subcutaneous injection of 100 µg/kg placebo for Navepegritide
  Arms: Placebo for Navepegritide

SUMMARY:
This trial is a Phase 2, multicenter, double-blind, randomized (ratio 2:1 TransCon CNP vs. placebo), placebo-controlled trial, designed to evaluate the safety, tolerability, and efficacy of 100 μg CNP/kg of Navepegritide (TransCon CNP) administered SC once-weekly for 52 weeks in infants with genetically verified heterozygous ACH, aged 0 to < 2 years at the time of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent by the parent(s)/caregiver(s) of the participant, and as required by the institutional review board/human research ethics committee/independent ethics committee (IRB/HREC/IEC).
* Male or female younger than 2 years of age at the time of randomization; or for open label sentinel participants, at the time of first administration of IMP.
* Clinical diagnosis of achondroplasia (ACH) with genetic confirmation of heterozygous genotype present during screening.
* Parent(s)/caregiver(s) willing to follow the protocol and instructions provided, including being able to administer weekly subcutaneous injections of trial treatment.
* Compliance to daily Vitamin D supplementation for infants aged 14 days to 1 year. All participants older than 1 year of age with serum 25-hydroxyvitamin D (25OHD) measured below lower limit of reference range at screening should start daily Vitamin D supplementation prior to randomization.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, ECG, imaging, and clinical laboratory tests performed during the screening period.

Exclusion Criteria:

* Known or suspected hypersensitivity to the investigational product or related products (trehalose, tris[hydroxymethyl]aminomethane, succinate, and polyethylene glycol [PEG]).
* Genetic confirmation of ACH homozygous genotype.
* Premature birth with gestational age < 32 weeks.
* Premature birth with gestational age 32 to 37 weeks, unless time from birth is > 6 months at the time of screening and the child is in good nutritional status, defined as gain in body weight expected for age and diagnosis of ACH, as determined by the Investigator and confirmed with the Medical Monitor.
* Anticipated, as assessed by Investigator and confirmed with Medical Monitor, to undergo surgical intervention during trial participation, including cervicomedullary decompression. Evaluation of immediate risk of requiring cervicomedullary decompression surgery will rely on the following assessments:

  * Physical examination (e.g., neurologic findings of clonus, opisthotonus, exaggerated reflexes, dilated facial veins)
  * Evidence of uncontrolled sleep apnea as confirmed by local standard of care assessment (e.g. polysomnography or simple sleep test) performed within 6 months prior to screening.
  * MRI performed at screening indicating presence of severe cervicomedullary compression (CMC) or spinal cord damage. Presence of abnormal MRI T2 signal intensity at and immediately above and below the cervicomedullary junction should be considered high risk for requiring surgery and the participant is not eligible for trial participation.

Common surgeries, such as insertion of grommets, adenoidectomy, tonsillectomy, or myringotomy tube placement are permitted during trial participation.

* Have a growth disorder or medical condition, other than ACH, resulting in short stature or abnormal growth as determined by the Investigator and confirmed with the Medical Monitor.
* Have received any dose of prescription medications and/or investigational medicinal product or device intended to affect stature, growth, or body proportionality (including human growth hormone or vosoritide) at any time.
* Requires or anticipated to require chronic (> 4 weeks) or repeated treatment (more than twice/year) with oral corticosteroids, or high-dose inhaled corticosteroids during trial participation.
* History or presence of injury or disease of the growth plate(s), other than ACH, affecting growth potential of long bones, including Salter-Harris fracture and recent bone-related surgery, as determined by Investigator and confirmed with the Medical Monitor.
* Have a clinically significant finding indicating abnormal cardiac function, including but not limited to:

  * Repaired or unrepaired coarctation.
  * Moderate or greater complexity congenital heart disease including tetralogy of Fallot, atrioventricular septal defects, truncus arteriosus, total anomalous pulmonary venous return, double outlet right ventricle, or single ventricle heart disease.
  * QTcF ≥ 450 msec on screening 12-lead ECG.
* History or presence of a condition impacting hemodynamic stability (such as autonomic dysfunction and orthostatic intolerance).
* History or presence of the following:

  * Chronic anemia.
  * Chronic renal insufficiency.
  * Chronic or recurrent illness that can affect hydration or volume status, including conditions associated with decreased nutritional intake or increased volume loss.
* History or presence of malignant disease.
* Any disease or condition that, in the opinion of the Investigator, may make the participant unlikely to fully complete the trial, not adhering to trial procedures, may confound interpretation of trial results, or may present undue risk from receiving trial treatment. This could include family situations, comorbid conditions, or medications that might impact safety or be considered confounding.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of Navepegritide | 52 weeks
  Incidence of treatment emergent adverse events (TEAEs)
To evaluate the effect of Navepegritide on growth | 52 weeks
  Change from baseline to 52 weeks in length/height Z-score

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S
Locations (17):
- United States (3):
  - Ascendis Investigational Site, Saint Paul, Minnesota
  - Ascendis Investigational Site, Houston, Texas
  - Ascendis Investigational Site, Madison, Wisconsin
- Ascendis Investigational Site, Parkville, Australia
- Ascendis Investigational Site, Linz, Austria
- Ascendis Investigational Site, Copenhagen, Denmark
- Ascendis Investigational Site, Helsinki, Finland
- Ascendis Investigational Site, Paris, France
- Germany (2):
  - Ascendis Investigational Site, Berlin
  - Ascendis Investigational Site, Cologne
- Ascendis Investigational Site, Dublin, Ireland
- Ascendis Investigational Site, Milan, Italy
- Ascendis Investigational Site, Auckland, New Zealand
- Ascendis Investigational Site, Oslo, Norway
- Ascendis Investigational Site, Coimbra, Portugal
- Ascendis Investigational Site, Stockholm, Sweden
- Ascendis Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No